CLINICAL TRIAL: NCT00540514
Title: A Randomized, Phase III Trial of ABI-007 and Carboplatin Compared With Taxol and Carboplatin as First-Line Therapy in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Albumin-bound Paclitaxel (ABI-007) for Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA031
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Non-Small Cell Lung Carcinoma
Keywords: Advanced Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Albumin-Bound Paclitaxel; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albumin-bound paclitaxel + Carboplatin (Experimental): Participants received albumin-bound paclitaxel (ABRAXANE®) 100 mg/m^2 administered as an intravenous infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle. Carboplatin was given at an Area Under the Curve (AUC) = 6 mg*min/mL on Day 1 only of each 21-day cycle, beginning immediately after the completion of albumin-bound paclitaxel administration. Participants could continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Albumin-bound paclitaxel; Drug: Carboplatin
- Paclitaxel + Carboplatin (Active Comparator): Participants received 200 mg/m^2 paclitaxel (Taxol®) administered by intravenous infusion followed by carboplatin at AUC = 6 mg*min/mL on Day 1 of a 21 day cycle. Participants could continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Albumin-bound paclitaxel — Administered by intravenous infusion.
  Other Names: ABI-007; ABRAXANE®; nab®-paclitaxel
  Arms: Albumin-bound paclitaxel + Carboplatin
Drug: Paclitaxel — Administered by intravenous infusion.
  Other Names: Taxol®
  Arms: Paclitaxel + Carboplatin
Drug: Carboplatin — Administered by intravenous infusion. Dosing was based on the Calvert formula: carboplatin dose (mg) = (Target AUC) x (glomerular filtration rate [GFR] + 25). For the purposes of this protocol, the GFR is considered to be equivalent to creatinine clearance (calculated by the method of Cockcroft and Gault, 1976).

SUMMARY:
The purpose of this study is to compare disease response of Albumin-bound paclitaxel (ABI-007) plus Carboplatin versus Taxol and Carboplatin as first-line therapy in patients with advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB or IV non-small cell lung cancer (NSCLC)
* Male or non-pregnant and non-lactating female, and equal or greater than age 18

  * If a female patient is of child-bearing potential, as evidence by regular menstrual periods, she must have a negative serum pregnancy test (beta human chorionic gonadotropin [βhCG]) documented within 72 hours of the first administration of study drug
  * If sexually active, the patient must agree to utilize contraception considered adequate and appropriate by the investigator
* No other current active malignancy
* Radiographically-documented measurable disease (defined by the presence of at least 1 radiographically documented measurable lesion)
* Patients must have received no prior chemotherapy for the treatment of metastatic disease. Adjuvant chemotherapy permitted providing cytotoxic chemotherapy was completed 12 months prior to starting the study
* Patient has the following blood counts at baseline:

  * Absolute neutrophil count (ANC) greater than or equal to 1.5x10^9/L
  * Platelets greater than or equal to 100x10^9/L
  * Hemoglobin (Hgb) greater than or equal to 9 g/dL
* Patient has the following blood chemistry levels at baseline:

  * Aspartate aminotransferase (SGOT), alanine aminotransferase (SGPT) less than or equal to 2.5 x upper limit of normal range (ULN) or less than or equal to 5.0 x ULN if liver metastases;
  * Total bilirubin less than or equal to ULN
  * Creatinine less than or equal to 1.5 mg/dL
* Expected survival of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patient or his/her legally authorized representative or guardian has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent form prior to participation in any study-related activities

Exclusion Criteria:

* Evidence of active brain metastases, including leptomeningeal involvement. Prior evidence of brain metastasis permitted only if treated and stable and off therapy for greater than or equal to 1 month
* The only evidence of disease is non-measurable
* Patient has pre-existing peripheral neuropathy of Grade 2, 3, or 4 (per Common Terminology Criteria for Adverse Events [CTCAE] Version 3).
* Patient received radiotherapy in the last 4 weeks, except if to a non-target lesion only. Prior radiation to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed
* Patient has a clinically significant concurrent illness
* Patient has received treatment with any investigational drug within the previous 4 weeks
* Patient has a history of allergy or hypersensitivity to any of the study drugs
* Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug
* Patient is enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2007-11-01 (Actual); Primary Completion 2009-10-01 (Actual); Study Completion 2013-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Socinski, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (37):
- United States (31):
  - Clearview Cancer Institute Oncology Specialties, P.C., Huntsville, Alabama
  - Genesis Cancer Center- Hot Springs, Hot Springs, Arkansas
  - Little Rock Hematology Oncology Associates, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Southwest Cancer Care, Escondido, California
  - Robert A. Moss, MD, FACP, Inc., Fountain Valley, California
  - Pacific Shores Medical Group, Long Beach, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Comprehensice Cancer Ctr., Palms Springs, California
  - Gulf Coast Oncology Associates, St. Petersburg, Florida
  - Lake County Oncology and Hematology, PA, Tavares, Florida
  - Phoebe Cancer Center, Albany, Georgia
  - Cancer Center of Kansas, Wichita, Kansas
  - Kentuckiana Cancer Institute, PLLC, Louisville, Kentucky
  - Mercy Hospital, Portland, Maine
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - St. Louis University, St Louis, Missouri
  - Essex Oncology of North Jersey, Belleville, New Jersey
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - St. Mary Medical Center- Oncology, Hematology PC, Langhorne, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dallas Oncology Consultants, PA, Duncanville, Texas
  - The Center for Cancers and Blood Disorders, Fort Worth, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - Tyler Hematology Oncology, Tyler, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Cancer Outreach Associates, PC, Abingdon, Virginia
- Canada (6):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - William Osler Health Centre, Brampton Clinic, Brampton, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University- Dept. of Oncology, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec

REFERENCES:
- [Background] Hirsh V. nab-paclitaxel for the management of patients with advanced non-small-cell lung cancer. Expert Rev Anticancer Ther. 2014 Feb;14(2):129-41. doi: 10.1586/14737140.2014.881719. PMID 24467217
- [Background] Langer CJ, Hirsh V, Ko A, Renschler MF, Socinski MA. Weekly nab-paclitaxel in combination with carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer: analysis of safety and efficacy in patients with renal impairment. Clin Lung Cancer. 2015 Mar;16(2):112-20. doi: 10.1016/j.cllc.2014.09.003. Epub 2014 Sep 30. PMID 25572008
- [Background] Langer CJ, Hirsh V, Okamoto I, Lin FJ, Wan Y, Whiting S, Ong TJ, Renschler MF, Botteman MF. Survival, quality-adjusted survival, and other clinical end points in older advanced non-small-cell lung cancer patients treated with albumin-bound paclitaxel. Br J Cancer. 2015 Jun 30;113(1):20-9. doi: 10.1038/bjc.2015.181. Epub 2015 Jun 2. PMID 26035702
- [Result] Socinski MA, Bondarenko I, Karaseva NA, Makhson AM, Vynnychenko I, Okamoto I, Hon JK, Hirsh V, Bhar P, Zhang H, Iglesias JL, Renschler MF. Weekly nab-paclitaxel in combination with carboplatin versus solvent-based paclitaxel plus carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer: final results of a phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2055-62. doi: 10.1200/JCO.2011.39.5848. Epub 2012 Apr 30. PMID 22547591
- [Result] Socinski MA, Langer CJ, Okamoto I, Hon JK, Hirsh V, Dakhil SR, Page RD, Orsini J, Zhang H, Renschler MF. Safety and efficacy of weekly nab(R)-paclitaxel in combination with carboplatin as first-line therapy in elderly patients with advanced non-small-cell lung cancer. Ann Oncol. 2013 Feb;24(2):314-321. doi: 10.1093/annonc/mds461. Epub 2012 Nov 2. PMID 23123509
- [Result] Satouchi M, Okamoto I, Sakai H, Yamamoto N, Ichinose Y, Ohmatsu H, Nogami N, Takeda K, Mitsudomi T, Kasahara K, Negoro S. Efficacy and safety of weekly nab-paclitaxel plus carboplatin in patients with advanced non-small cell lung cancer. Lung Cancer. 2013 Jul;81(1):97-101. doi: 10.1016/j.lungcan.2013.02.020. Epub 2013 Mar 30. PMID 23545279
- [Result] Socinski MA, Okamoto I, Hon JK, Hirsh V, Dakhil SR, Page RD, Orsini J, Yamamoto N, Zhang H, Renschler MF. Safety and efficacy analysis by histology of weekly nab-paclitaxel in combination with carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer. Ann Oncol. 2013 Sep;24(9):2390-6. doi: 10.1093/annonc/mdt235. Epub 2013 Jul 10. PMID 23842283
- [Result] Hirsh V, Okamoto I, Hon JK, Page RD, Orsini J, Sakai H, Zhang H, Renschler MF, Socinski MA. Patient-reported neuropathy and taxane-associated symptoms in a phase 3 trial of nab-paclitaxel plus carboplatin versus solvent-based paclitaxel plus carboplatin for advanced non-small-cell lung cancer. J Thorac Oncol. 2014 Jan;9(1):83-90. doi: 10.1097/JTO.0000000000000011. PMID 24346096
- [Derived] Loureiro H, Kolben TM, Kiermaier A, Ruttinger D, Ahmidi N, Becker T, Bauer-Mehren A. Correlation Between Early Trends of a Prognostic Biomarker and Overall Survival in Non-Small-Cell Lung Cancer Clinical Trials. JCO Clin Cancer Inform. 2023 Sep;7:e2300062. doi: 10.1200/CCI.23.00062. PMID 37922432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible patients were randomized on Day 1 in a 1:1 ratio into 1 of 2 treatment arms and were required to start treatment within 7 days of randomization. The data below represent a cut-off of 31 January 2011. One patient was randomized twice and not included in the Intent-to-treat population.
Groups:
- Albumin-bound Paclitaxel + Carboplatin: Participants received albumin-bound paclitaxel (ABRAXANE®) 100 mg/m^2 administered as an intravenous (IV) infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle. Carboplatin was given at an Area Under the Curve (AUC) = 6 mg*min/mL on Day 1 only of each 21-day cycle, beginning immediately after the completion of albumin-bound paclitaxel administration. Participants could continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.
- Paclitaxel + Carboplatin: Participants received 200 mg/m^2 paclitaxel (Taxol®) administered by intravenous infusion followed by carboplatin at AUC = 6 mg*min/mL on Day 1 of a 21-day cycle. Participants could continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Started | 521 (Intent-to-treat Population: all randomized patients regardless of treatment received.) | 531 (Intent-to-treat Population: all randomized patients regardless of treatment received.)
Treated | 514 | 524
Biomarker Population | 35 | 36
Completed | 275 (Completed defined as discontinuation due to progressive disease) | 265 (Completed defined as discontinuation due to progressive disease)
Not Completed | 246 | 266
Not completed — Still on treatment | 3 | 0
Not completed — Unacceptable Toxicity | 61 | 62
Not completed — Adverse Event | 20 | 24
Not completed — Physician Decision | 86 | 99
Not completed — Protocol Deviation | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 65 | 67
Not completed — Excluded prior to treatment | 7 | 7
Not completed — Paclitaxel not available | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Albumin-bound Paclitaxel + Carboplatin: Participants received albumin-bound paclitaxel 100 mg/m^2 administered as an intravenous infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle. Carboplatin was given at an Area Under the Curve (AUC) = 6 mg*min/mL on Day 1 only of each 21-day cycle, beginning immediately after the completion of albumin-bound paclitaxel administration. Participants could continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.
- Paclitaxel + Carboplatin: Participants received 200 mg/m^2 paclitaxel administered by intravenous infusion followed by carboplatin at AUC = 6 mg*min/mL on Day 1 of a 21-day cycle. Participants could continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 521 | 531 | 1052
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.14) | 59.7 (9.53) | 59.6 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 134 | 263
  Male | 392 | 397 | 789
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 79 | 80 | 159
  Black, of African Heritage | 12 | 8 | 20
  North American Indian or Alaska Native | 1 | 0 | 1
  White, Non Hispanic and Non Latino | 416 | 433 | 849
  White, Hispanic or Latino | 11 | 5 | 16
  Other | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 63 | 58 | 121
  Canada | 21 | 23 | 44
  Australia | 5 | 9 | 14
  Japan | 74 | 75 | 149
  Russian Federation | 238 | 231 | 469
  Ukraine | 120 | 135 | 255
Smoking status [Number; unit: participants]
  Never smoked | 137 | 144 | 281
  Smoked and quit smoking | 168 | 148 | 316
  Smoked and currently smokes | 214 | 234 | 448
  Missing | 2 | 5 | 7
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A scale used to assess the progress of disease in a patient, how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  participants
    0 (Fully active) | 133 | 113 | 246
    1 (Restrictive but ambulatory) | 385 | 416 | 801
    2 (Ambulatory but unable to work) | 3 | 2 | 5
Time from Primary Diagnosis to Study Entry [Mean (Standard Deviation); unit: months] | 4.3 (17.12) | 4.3 (16.09) | 4.3 (16.60)
Stage at Primary Diagnosis [Number; unit: participants] — I: The tumor has not spread outside the chest or to the lymph nodes.
  II: A tumor that may have spread to local lymph nodes, but has not spread further.
  IIIa: A tumor of any size, cancer cells are found in the lymph nodes near the lungs and bronchi and in the lymph nodes between the lungs on the same side of the chest.
  IIIb: Any size tumor that has spread to distant lymph nodes, or invaded other structures in the chest such as the heart or esophagus, or a tumor with a malignant pleural effusion.
  IV - The cancer has spread to another part of the body, including the opposite lung.
  participants
    I | 16 | 20 | 36
    II | 18 | 24 | 42
    IIIa | 22 | 24 | 46
    IIIb | 135 | 116 | 251
    IV | 325 | 344 | 669
    Unknown | 5 | 3 | 8
Anatomic Site of Primary Diagnosis [Number; unit: participants]
  Lung | 480 | 499 | 979
  Other | 41 | 32 | 73
Histology of Primary Diagnosis [Number; unit: participants]
  Carcinoma/ Adenocarcinoma | 254 | 264 | 518
  Squamous Cell Carcinoma | 229 | 221 | 450
  Large Cell Carcinoma | 9 | 13 | 22
  Other | 29 | 33 | 62
Time from 1st Documented Metastasis/Relapse to Study Entry [Mean (Standard Deviation); unit: months] | 0.9 (2.11) | 0.8 (1.25) | 0.9 (1.73)
Stage at Randomization [Number; unit: participants]
  IIIb | 108 | 110 | 218
  IV | 413 | 421 | 834

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Objective Confirmed Complete Response or Partial Response by Blinded Radiology Assessment
Description: Antitumor response was defined as the percentage of participants who achieved an objective response (Confirmed Response [CR] or Partial Response [PR]), confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. Response was based on the blinded radiological review using Response Evaluation Criteria in Solid Tumors (RECIST) response guidelines, Version 1.0.
  A complete response was defined as a disappearance of all target and non-target lesions and no new lesions.
  Partial response was defined as ≥ 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD, and the persistence of one or more non-target lesions not qualifying for CR or Progressive Disease (the "unequivocal progression" of existing non-target lesion(s) or appearance of one or more new lesions).
Time Frame: Objective response was evaluated every 6 weeks until progression or new anti-cancer therapy initiation, up to 22 months.
Population: The intent-to-treat population which includes all randomized patients regardless of whether the patient received any study drug or had any efficacy assessments collected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 521 | 531
percentage of participants | 33 [28.6 to 36.7] | 25 [21.2 to 28.5]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; The null hypothesis is that the albumin-bound paclitaxel/carboplatin regimen response rate (PA) is equal to that of the paclitaxel (Taxol)/carboplatin regimen (PT). Superiority of albumin-bound paclitaxel/carboplatin to paclitaxel/carboplatin will be established if the lower bound of the 95.1% CI of the response rate ratio is > 1.0; Test type: Superiority or Other; p = 0.005, Chi-squared — Statistical significance defined as P-value < 0.049; Response Rate Ratio = 1.313, 95.1% CI 2-sided [1.082 to 1.593] — Response rate ratio = PA/PT. A response rate ratio > 1 favors the albumin-bound paclitaxel/carboplatin arm of the study

2. Secondary Outcome: Progression-free Survival by Blinded Radiology Assessment
Description: Progression free survival time was defined as the time from the day of randomization to the start of disease progression or death (any cause), whichever occurred first, based on the blinded radiological review response assessment. Progressive disease was defined as a ≥ 20% increase in the SLD of target lesions, taking as reference the nadir SLD recorded since the treatment started, or the presence of one or more new lesions, or the "unequivocal progression" of existing non-target lesion(s) or appearance of one or more new lesion(s).
  Participants who did not have disease progression or had not died were censored at the last visit they were documented as progression free. If palliative radiotherapy or surgery at lesion sites occurred, the participant was censored at the last date without documented progression prior to radiotherapy or surgery. In follow-up, participants who began new therapy prior to progression were censored at the last documented date as progression-free.
Time Frame: Assessed every 6 weeks until progression or death, up to 38 months
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 521 | 531
months | 6.3 [5.6 to 7.0] | 5.8 [5.6 to 6.7]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.214, Log Rank — P-value is based on a stratified log rank test stratified by geographic region (North America/Australia, Eastern Europe, or Asia/Pacific) and histology of primary diagnosis (squamous cell carcinoma, adenocarcinoma, or other carcinoma); Hazard Ratio (HR) = 0.902, 95.1% CI 2-sided [0.767 to 1.060] — Hazard ratio (albumin-bound paclitaxel/carboplatin to paclitaxel/carboplatin) <1 favors the albumin-bound paclitaxel/carboplatin group

3. Secondary Outcome: Overall Participant Survival
Description: Overall survival was defined as the time from the day of randomization to participant death (due to any cause), as assessed by post study follow-up performed monthly for 6 months and every 3 months thereafter for 12 months. All participants who were lost to the follow-up prior to the end of the trial or who completed the 18 month follow up phase were censored at last known time the participant was alive.
Time Frame: Up to 38 months
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 521 | 531
months | 12.1 [10.8 to 12.9] | 11.2 [10.3 to 12.6]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.271, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.922, 95.1% CI 2-sided [0.797 to 1.066] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With Controlled Disease
Description: Controlled disease was defined as the percentage of participants with stable disease for ≥ 16 weeks or confirmed complete or partial overall response, based on blinded radiological assessment. Stable disease was defined as neither sufficient shrinkage of target lesions to qualify for Partial Response, nor sufficient increase to qualify for Progressive Disease, or the persistence of one or more non-target lesions not qualifying for Complete Response or Progressive Disease.
Time Frame: Assessed every 6 weeks, up to 22 months
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 521 | 531
percentage of participants | 53 [48.3 to 56.9] | 49 [44.7 to 53.2]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.239, Chi-squared; Response Rate Ratio = 1.074, 95% CI 2-sided [0.953 to 1.210]

5. Secondary Outcome: Duration of Response in Responding Patients
Description: Duration of response was assessed by progression free survival for participants who achieved a confirmed complete response or partial response based on blinded radiological assessment.
Time Frame: Assessed every 6 weeks, up to 38 months
Population: Intent-to-treat patients with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 170 | 132
months | 9.6 [8.3 to 10.8] | 9.5 [8.1 to 11.0]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.551, Log Rank — P-value is based on a stratified log rank test stratified by geographic region (North America/Australia, Eastern Europe, or Asia/Pacific) and histology of primary diagnosis (Squamous cell carcinoma or Non squamous cell carcinoma); Hazard Ratio (HR) = 0.901, 95% CI 2-sided [0.652 to 1.244] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A Treatment-emergent AE was any AE that began or worsened in grade after the start of study drug through 30 days after the last dose of study drug or end of study whichever is later. Treatment related toxicity was one considered by the investigator to be possibly, probably or definitely related to study drug. AEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 on the following scale: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death. A serious adverse event (SAE) is any untoward medical occurrence at any dose that: is fatal or life-threatening; results in persistent or significant disability or incapacity; requires or prolongs in-patient hospitalization; is a congenital anomaly/birth defect in the offspring of a patient; and conditions not included in the above that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Up to 38 months
Population: Treated population
Measure: Number; unit: participants
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 514 | 524
participants
  At least 1 AE | 483 | 504
  At least 1 grade 3 or higher AE | 360 | 355
  At least 1 treatment-related AE | 469 | 481
  At least 1 treatment-related grade 3 or higher AE | 321 | 315
  At least 1 serious AE | 93 | 80
  At least 1 treatment-related serious AE | 37 | 30
  At least 1 AE with taxane permanently discontinued | 80 | 84
  At least 1 AE with action of taxane dosage reduced | 237 | 120
  At least 1 AE with action of taxane interrupted | 0 | 5
  At least 1 AE with action of taxane delayed | 365 | 214

7. Secondary Outcome: Pharmacokinetic (PK) Parameters
Time Frame: Blood samples for PK analyses were taken during Cycle 1 at 0.25, 3.5 and 24 hours post-infusion.
Population: Patients randomized to receive albumin-bound paclitaxel/carboplatin treatment in Canada, Russia, Ukraine and United States had the option to participate in sparse PK sampling in this study. Only 15 participants consented to participate, an insufficient number to support the planned population PK analysis hence these analyses were not performed.
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: SPARC Status and Correlation With Overall Survival
Description: The expression and cellular distribution of Secreted Protein Acidic and Rich in cysteine (SPARC) in biopsies of lung tumor was examined by immunohistochemistry using a 2 antibody system by an approved central laboratory and analyzed by 2 pathologists. The following tissue components were scored: tumor cells, fibroblasts, inflammatory cells, acellular stroma/matrix, and blood vessels.
  To classify participants into "high-SPARC" and "low-SPARC" groups, an average z-score was calculated across variables and classified "high-SPARC" (average z-scores ≥0) and "low-SPARC" (average z-scores <0) groups.
  SPARC status was then correlated with overall survival (the time from the day of randomization to participant death due to any cause).
Time Frame: Archival tissue samples were used for SPARC analysis. Survival was assessed for up to 38 months.
Population: SPARC biomarker Population
Measure: Number; unit: participants
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 35 | 36
participants
  High-SPARC | 17 [3.3 to 23.1] | 22 [2.3 to 28.0]
  Low-SPARC | 18 [3.7 to 24.9] | 14 [4.7 to 22.3]
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel + Carboplatin vs Paclitaxel + Carboplatin; SPARC correlation with overall survival for the overall SPARC population; Test type: Superiority or Other; p = 0.302, Univariate Cox regression

9. Other Pre Specified Outcome: Percentage of Participants Who Achieved an Objective Confirmed Complete Response or Partial Response by Blinded Radiology Assessment, by Histology
Description: Antitumor response was defined as the percentage of participants who achieved an objective response (Confirmed Response [CR] or Partial Response [PR]), confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. Response was based on the blinded radiological review using Response Evaluation Criteria in Solid Tumors (RECIST) response guidelines, Version 1.0.
  A complete response was defined as a disappearance of all target and non-target lesions and no new lesions.
  Partial response was defined as ≥ 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD, and the persistence of one or more non-target lesions not qualifying for CR or Progressive Disease (the "unequivocal progression" of existing non-target lesion(s) or appearance of one or more new lesions).
  Histology was determined at the time of primary diagnosis.
Time Frame: Objective response was evaluated every 6 weeks until progression or new anti-cancer therapy initiation, up to 22 months.
Population: The intent-to-treat population. N indicates the number of participants in each histology category for each treatment arm respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 521 | 531
percentage of participants
  Carcinoma/Adenocarcinoma [254, 264] | 26 | 27
  Squamous Cell Carcinoma [229, 221] | 41 | 24
  Large Cell Carcinoma [N=9, 13] | 33 | 15
  Other [N=29, 33] | 24 | 15
Statistical Analysis 1: Comparison: Albumin-bound Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.036, Regression, Logistic — A nonsignificant interaction P-value (ie, p-value ≥ 0.100) indicates the treatment regimen effect was consistent within a prognostic factor; Logistic regression model with effects for treatment regimen, prognostic factor (histology), and treatment regimen by prognostic factor interaction

10. Other Pre Specified Outcome: Maximal Degree of Anemia Based on Clinical Laboratory Values for Hemoglobin
Description: The maximal degree of anemia (and myelosuppression) was assessed by the overall nadir of hemoglobin levels based on clinical laboratory measurements graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
Time Frame: 38 months
Population: Treated population where laboratory data were available.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Albumin-bound Paclitaxel + Carboplatin: Participants received albumin-bound paclitaxel 100 mg/m^2 administered as an intravenous (IV) infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle. Carboplatin was given at an Area Under the Curve (AUC) = 6 mg*min/mL on Day 1 only of each 21-day cycle, beginning immediately after the completion of albumin-bound paclitaxel administration. Participants could continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 508 | 514
g/L | 90.0 (17.19) | 103.9 (16.90)

11. Other Pre Specified Outcome: Maximal Degree of Neutropenia Based on Clinical Laboratory Values of Absolute Neutrophil Count
Description: The maximal degree of neutropenia (and myelosuppression) was assessed by the overall nadir of absolute neutrophil count (ANC) based on clinical laboratory measurements graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
Time Frame: 38 months
Population: Treated population where laboratory data were available.
Measure: Mean (Standard Deviation); unit: × 10^9/L
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 508 | 513
× 10^9/L | 1.39 (1.721) | 1.26 (1.366)

12. Other Pre Specified Outcome: Maximal Degree of Thrombocytopenia Based on Clinical Laboratory Values of Platelet Count
Description: The maximal degree of thrombocytopenia (and myelosuppression) was assessed by the overall nadir of platelet count based on clinical laboratory measurements graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
Time Frame: 38 months
Population: Treated population where laboratory data were available.
Measure: Mean (Standard Deviation); unit: × 10^9/L
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 508 | 513
× 10^9/L | 114.9 (82.13) | 136.6 (81.91)

13. Other Pre Specified Outcome: Time to Improvement of ≥ Grade 3 Treatment Related Peripheral Neuropathy
Description: Peripheral neuropathy was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 on the following scale: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death.
  Improvement in peripheral neuropathy was evaluated as:
  * Time to improvement of grade 3 or higher peripheral neuropathy by at least one grade;
  * Time to improvement of grade 3 or higher peripheral neuropathy to grade 1.
  Time to improvement was defined as the time from the first occurrence of grade 3 or higher treatment related neuropathy to improvement, as defined. Participants not experiencing improvement were censored at the last time the participant was evaluated for adverse events.
Time Frame: 38 months
Population: Treated population with ≥ grade 3 treatment-related peripheral neuropathy.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 17 | 62
days
  Improvement by ≥1 grade | 24.0 [15.0 to NA] — Maximum confidence interval limit not estimable due to low number of events. | 26.0 [15.0 to 38.0]
  Improvement to grade 1 | 38.0 [19.0 to NA] — Maximum confidence interval limit not estimable due to low number of events. | 104.0 [40.0 to 169.0]

ADVERSE EVENTS:
Time Frame: Up to 38 months
Arm/Group | Albumin-bound Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 93/514 | 80/524
Other Adverse Events (participants affected / at risk) | 483/514 | 499/524
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin-bound Paclitaxel + Carboplatin (N=514) | Paclitaxel + Carboplatin (N=524)
Anaemia (Blood and lymphatic system disorders) | 19 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 14 | 11
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Injection site abscess (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Convulsion (Nervous system disorders) | 2 | 1
Spinal cord compression (Nervous system disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 1 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Disease progression (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Influenza serology (Investigations) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin-bound Paclitaxel + Carboplatin (N=514) | Paclitaxel + Carboplatin (N=524)
Neutropenia (Blood and lymphatic system disorders) | 260 | 250
Anaemia (Blood and lymphatic system disorders) | 225 | 109
Thrombocytopenia (Blood and lymphatic system disorders) | 208 | 122
Leukopenia (Blood and lymphatic system disorders) | 97 | 91
Alopecia (Skin and subcutaneous tissue disorders) | 287 | 312
Rash (Skin and subcutaneous tissue disorders) | 50 | 43
Peripheral sensory neuropathy (Nervous system disorders) | 136 | 209
Neuropathy peripheral (Nervous system disorders) | 104 | 118
Dysgeusia (Nervous system disorders) | 36 | 33
Headache (Nervous system disorders) | 36 | 23
Dizziness (Nervous system disorders) | 31 | 20
Fatigue (General disorders) | 126 | 120
Asthenia (General disorders) | 83 | 75
Oedema peripheral (General disorders) | 53 | 21
Pyrexia (General disorders) | 48 | 41
Chest pain (General disorders) | 27 | 20
Nausea (Gastrointestinal disorders) | 140 | 130
Constipation (Gastrointestinal disorders) | 84 | 67
Vomiting (Gastrointestinal disorders) | 63 | 63
Stomatitis (Gastrointestinal disorders) | 29 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 | 59
Diarrhoea (Gastrointestinal disorders) | 75 | 58
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 38
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 36 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 21 | 27
White blood cell count decreased (Investigations) | 60 | 64
Haemoglobin decreased (Investigations) | 56 | 34
Neutrophil count decreased (Investigations) | 55 | 58
Alanine aminotransferase increased (Investigations) | 46 | 44
Weight decreased (Investigations) | 43 | 33
Aspartate aminotransferase increased (Investigations) | 42 | 31
Platelet count decreased (Investigations) | 34 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 65 | 129
Myalgia (Musculoskeletal and connective tissue disorders) | 50 | 97
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 28
Decreased appetite (Metabolism and nutrition disorders) | 89 | 96
Insomnia (Psychiatric disorders) | 28 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the results of its findings if a multicenter publication is not forthcoming within 18 months after study completion. Institution shall provide Celgene with a copy of the papers prior to their submission; Celgene shall complete its review within 60 days after receipt. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of patentable material.